CLINICAL TRIAL: NCT01791075
Title: Prospective Randomized Study Comparing Endothelial Cell Loss Using the Tan EndoGlide With the Endoserter for Insertion of the Donor Graft in Descemets Stripping Endothelial Keratoplasty (DSAEK)
Brief Title: Comparing Endoglide to Endoserter for DSAEK Graft Insertion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB 10-0631-B
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Fuch's Endothelial Dystrophy; Bullous Keratopathy, Unspecified Eye
Keywords: DSAEK; Tan Endoglide; Endosaver/Endoserter
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tan Endoglide (Active Comparator): Patients assigned to this arm will have their endothelial donor graft injected into the anterior chamber using the Tan Endoglide.
  Interventions: Device: Tan Endoglide
- Endosaver/serter (Active Comparator): Patients assigned to this arm will have their endothelial donor graft injected into the anterior chamber using the Endosaver/serter injector.
  Interventions: Device: Endosaver

INTERVENTIONS:
Device: Tan Endoglide — Patients assigned to this intervention will have their endothelial donor graft injected into the anterior chamber using the Tan Endoglide
  Arms: Tan Endoglide
Device: Endosaver — Patients assigned to this intervention will have their endothelial donor graft injected into the anterior chamber using the Tan Endoglide
  Other Names: Endoserter
  Arms: Endosaver/serter

SUMMARY:
The purpose of this study is to compare the Tan EndoGlide with the new Endoserter injector in terms of damage to the donor corneal endothelium by comparing the endothelial cell loss at 1 month, 3 months, 6 months, and 1 year post DSAEK (Descemet's Stripping Automated Endothelial Keratoplasty)surgery. There is no data comparing this two injectors.

DETAILED DESCRIPTION:
Descemet's stripping automated endothelial keratoplasty (DSAEK) is a widely performed method of corneal transplantation. It is now considered the standard of care for the treatment of endothelial cell dysfunction. The advantages of this technique include faster visual rehabilitation, decreased risk of allograft rejection, preservation of corneal tectonic strength, stable refraction, reduced irregular astigmatism, and less suture complications.

The standard of care at the Toronto Western Hospital for Dr. Rootman's and Dr. Slomovic's patients with corneal endothelial disease is to perform DSAEK surgery with the Tan Endoglide for insertion of the donor graft. Other surgeons at Toronto Western Hospital use either Busin glide or specifically designed forceps for insertion of the donor graft as part of the standard of care. Still others have advocated the use of the suture pull-through technique.

There is significant disagreement in the literature regarding the DSAEK insertion technique that best preserves the donor endothelium. Some investigators report better results with a forceps or sutures, and others caution against any folding. The less traumatic the insertion to the endothelium, the better the long term survival of the corneal transplant. In addition, surgeons also debate whether large- or small-incision DSAEK is better for the graft's long-term viability, its propensity for postoperative dislocation, and the ease of insertion in the OR. The proposed advantages of the Tan EndoGlide include consistent and reliable delivery of the corneal donor through a small incision with minimal endothelial loss. The advantages of a small-incision DSAEK are, that it provides a more stable wound postoperatively, sutureless surgery, speed, and convenience for combining the procedure with standard phacoemulsification. Balancing the attractiveness of small-incision DSAEK with the concern for endothelial injury from donor folding and forceps compression, the Endosaver (Ocular Systems, Inc., Winston-Salem, NC) a novel DSAEK injector device, has been recently introduced. It allows the surgeon to insert unfolded tissue without a forceps through a 4-mm clear corneal incision.

Both devices have been approved for use by Health Canada as a Class 1 device (http://www.angioedupro.com/Sharpoint/index.php?seek=394).

Recently, the results of a randomised prospective study being conducted by Dr. D. Tan (inventor of the Tan EndoGlide) were published. In this study the effect on endothelial cell counts using the Tan EndoGlide has been evaluated. The investigators report a 15.6% of endothelial cell loss 12 months after DSAEK surgery. There are no published studies regarding the Endosaver injector, nevertheless, preliminary results indicate poorer outcome (30% cell loss after one month). No study comparing the two devices in regard to endothelial cell loss was reported so far.

The purpose of this study is to compare the Tan EndoGlide with the new Endosaver injector in terms of damage to the donor corneal endothelium by comparing the endothelial cell loss at 1 month, 3 months, 6 months, and 1 year postoperatively. Our study would involve prospectively examining a total of 42 subjects (21 eyes with the Tan EndoGlide and 21 eyes with the Endosaver injector) and compare endothelial cell loss and visual outcomes between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with corneal decompensation requiring DSAEK with or without cataract surgery for visual rehabilitation.
* Clinical diagnosis include endothelial cell dysfunction secondary to Fuchs endothelial dystrophy, pseudophakic or aphakic bullous keratopathy, failed penetrating keratoplasty or DSAEK, iridocorneal endothelial syndrome or trauma.
* Ability to understand the nature of the procedure and give full informed consent.
* Patients who are able to comply with the standard DSAEK follow-up protocol at the Toronto Western Hospital.

Exclusion Criteria:

* Patients with late stage corneal decompensation with stromal scarring unsuitable for DSAEK and therefore requiring penetrating keratoplasty.
* Patients with complex anterior segment pathology precluding successful DSAEK procedure.
* Patients not giving full informed consent to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Endothelial cell count after 6 months and 12 months | 6,12 months post op
  The patients will be evaluated for endothelial cell loss 6 and 12 post surgery

SECONDARY OUTCOMES:
Visual acuity | 1 month and 3,6,12 months post surgery
  The patients will be evaluated for Visual acuity stability/improvement at the previous mentioned intervals.

CONTACTS AND LOCATIONS:
Overall Officials: David S. Rootman, MD, Principal Investigator — TWH - UHN
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada